CLINICAL TRIAL: NCT02703792
Title: Enhanced Care Home Outcomes (ECHO): An Evaluation of the Experiences of Staff and Stakeholders Working With an Integrated Care Home Support Service (CHSS)
Brief Title: Enhanced Care Home Outcomes: A Qualitative Study
Acronym: ECHO
Status: Completed | Type: Observational
Sponsor: Oxford Health NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 1163
Record Dates: First submitted 2016-02-24; First posted 2016-03-09 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-04

CONDITIONS: Staff Attitude

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Care home staff: Care home staff working in the homes in the top 10% of service use of the 102 participating homes referring to the Care Home Support Service
- NHS staff: GPs supporting residents living in the top 10% of service use of the 102 participating homes referring to the Care Home Support Service
- Service user representatives: Service or carers of an older person with dementia attending and Age UK carers group
- Relatives of residents: Relatives of residents living in the top 10% of service use of the 102 participating homes referring to the Care Home Support Service

SUMMARY:
This qualitative study uses focus group methodology and purposive sampling with the aim of obtaining views of Care Home Support Service staff and other stakeholders about their experiences of a redesigned National Health Service (NHS) Care Home Support Service. Individual stakeholder focus groups will be conducted with General Practitioners (GP), care home staff, relatives of residents in care homes, service-user representatives (Total N=32, across 4 focus groups). This study forms part of a larger evaluation of the CHSS service; service improvement workshops will be conducted with Oxford Health NHS Care Home Support Service, Community Nursing and Community Mental Health staff that are working in the 102 participating homes. Each participant who consents will take part in a focus group to explore their experiences of a redesigned NHS care home support service. Participants will be involved in the study for up to six months from gaining informed consent until last contact with the research team when a summary of the research will be sent. The data will be analysed using thematic analysis and applied with the Reach, Effectiveness, Adoption, Implementation and Maintenance (RE-AIM) framework.

DETAILED DESCRIPTION:
There are currently 800 000 people in the United Kingdom (UK) living with dementia and this is predicted to grow to 1 million people by 2021. Studies suggest that 250 000 of people with dementia reside in care homes. Reports such as the National Dementia Strategy and subsequent government initiatives, such as the Dementia Challenge and the Prime Minister's Challenge on Dementia 2020 have helped the nation focus on provision of services for people with dementia. Further, our media remind us that the quality of care being delivered in care homes needs significant improvement. With an ageing population effective, safe, good quality care for our older people is paramount.

A high proportion of people in care homes have dementia and many have co-existing physical health problems and/or additional mental health needs. An integrated Care Home Support Service (CHSS) delivers care and treatment of both physical and mental health problems at an early stage of development. This integrated service combines two approaches which have been shown to be effective in randomised control trials and open studies in a stepped care model. Evidence suggests it is feasible to implement some elements of such approaches into a specialist mental health NHS context. However, no widespread implementation of this combined approach had been undertaken in an NHS context until the integration of this Care Home Support Service.

Evaluating the implementation of health care initiatives is crucial in determining their impact and sustainability in a routine NHS setting. This qualitative evaluation is part of a broader evaluation of the service. Focus groups and service improvement workshops will be conducted with NHS staff and other stakeholders. The data will be analysed using thematic analysis and applied to the RE-AIM framework to:

* Provide valuable information from NHS staff and stakeholders regarding the impact and sustainability of this model.
* Explore key factors to consider when integrating physical and mental health services.
* Increase understanding of the potential barriers and facilitators of integrating evidence-based practice into a routine NHS setting.

On completion of the research the findings of the study will be disseminated to research participants and health professionals to support learning and best practice both locally and nationally.

ELIGIBILITY:
Inclusion Criteria:

* Care home staff working in the homes in the top 10% of service use of the 102 participating homes referring to the Care Home Support Service*
* Relatives of residents living in the top 10% of service use of the 102 participating homes referring to the Care Home Support Service*
* GPs supporting residents living in the top 10% of service use of the 102 participating homes referring to the Care Home Support Service*
* Service user representatives from Age UK carer groups
* Note: * Sampling GPs, care staff and relatives through the top 10% of care homes referring to and using services of the care home support service will ensure that they have adequate awareness of the care home support team to contribute to the focus group discussion.

Exclusion Criteria:

* Not fluent in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Staff and relatives of service users
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2016-03; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Themes derived from a thematic analysis of staffs attitudes to the implementation an integrated care home in-reach team. | 1.5 hour focus group

CONTACTS AND LOCATIONS:
Locations (1):
- Department of psychological services, Fulbrook centre, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ballard C, Brown R, Fossey J, Douglas S, Bradley P, Hancock J, James IA, Juszczak E, Bentham P, Burns A, Lindesay J, Jacoby R, O'Brien J, Bullock R, Johnson T, Holmes C, Howard R. Brief psychosocial therapy for the treatment of agitation in Alzheimer disease (the CALM-AD trial). Am J Geriatr Psychiatry. 2009 Sep;17(9):726-33. doi: 10.1097/JGP.0b013e3181b0f8c0. PMID 19700946
- [Background] Ballard C, Orrell M, YongZhong S, Moniz-Cook E, Stafford J, Whittaker R, Woods B, Corbett A, Garrod L, Khan Z, Woodward-Carlton B, Wenborn J, Fossey J. Impact of Antipsychotic Review and Nonpharmacological Intervention on Antipsychotic Use, Neuropsychiatric Symptoms, and Mortality in People With Dementia Living in Nursing Homes: A Factorial Cluster-Randomized Controlled Trial by the Well-Being and Health for People With Dementia (WHELD) Program. Am J Psychiatry. 2016 Mar 1;173(3):252-62. doi: 10.1176/appi.ajp.2015.15010130. Epub 2015 Nov 20. PMID 26585409
- [Background] Brooker DJ, Latham I, Evans SC, Jacobson N, Perry W, Bray J, Ballard C, Fossey J, Pickett J. FITS into practice: translating research into practice in reducing the use of anti-psychotic medication for people with dementia living in care homes. Aging Ment Health. 2016 Jul;20(7):709-18. doi: 10.1080/13607863.2015.1063102. Epub 2015 Jul 13. PMID 26167720
- [Background] Fossey J, Ballard C, Juszczak E, James I, Alder N, Jacoby R, Howard R. Effect of enhanced psychosocial care on antipsychotic use in nursing home residents with severe dementia: cluster randomised trial. BMJ. 2006 Apr 1;332(7544):756-61. doi: 10.1136/bmj.38782.575868.7C. Epub 2006 Mar 16. PMID 16543297
- [Background] Glasgow RE, Vogt TM, Boles SM. Evaluating the public health impact of health promotion interventions: the RE-AIM framework. Am J Public Health. 1999 Sep;89(9):1322-7. doi: 10.2105/ajph.89.9.1322. PMID 10474547
- See also: Alzheimer's Society (2012). Dementia 2012: A National challenge report — https://www.alzheimers.org.uk/site/scripts/download_info.php?downloadID=821
- See also: Department of Health (2009). Living well with dementia: A national dementia strategy. Leeds: Author. — https://www.gov.uk/government/uploads/system/uploads/attachment_data/file/168220/dh_094051.pdf
- See also: Department of Health (2012). Prime Minister's challenge on dementia: Delivering major improvements in dementia care and research by 2015. Leeds: Author — https://www.gov.uk/government/uploads/system/uploads/attachment_data/file/215101/dh_133176.pdf
- See also: Department of Health (2015). Prime Minister's challenge on dementia 2020. Leeds: Author — https://www.gov.uk/government/uploads/system/uploads/attachment_data/file/414344/pm-dementia2020.pdf
- See also: James I. A. (2011). Understanding Behaviour in Dementia that Challenges. London: Jessica Kingsley Press — http://www.jkp.com/uk/understanding-behaviour-in-dementia-that-challenges.html
- See also: Knapp, M. Comas-Herrera, A. Somani, A. & Banerjee, S. (2007) Dementia:International Comparisons Personal Social Services Research unit, London — http://eprints.lse.ac.uk/3353/1/dementia_international_comparison_(published_version).pdf
- See also: Stone, C., Fossey,J., Broad, A. (2016) The Oxfordshire Integrated Care Home Support Service : New developments to address the health and well-being of people with dementia in care homes. The Psychology of Older People: The FPOP Bulletin. 133(Jan) 58-65. — http://shop.bps.org.uk/publications/publication-by-series/psige-newsletter/fpop-bulletin-133-january-2016.html